CLINICAL TRIAL: NCT03584789
Title: De-Implementing Opioid Use and Implementing Optimal Pain Management Following Dental Extractions
Brief Title: De-Implementing Opioids for Dental Extractions
Acronym: DIODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Friends Research Institute, Inc. (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A17-013; U01DE027441 (NIH)
Record Dates: First submitted 2018-06-08; First posted 2018-07-12 (Actual); Results first posted 2022-07-19 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-05

CONDITIONS: Tooth Extraction
Keywords: Decision Support Systems, Clinical; Pain Management; Analgesics
MeSH Terms: conditions — Agnosia | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Practice (No Intervention): The patients in this arm were part of usual care with their dental provider.
- Clinical Decision Support (Experimental): A clinical decision support system designed to assist dentists in providing optimal pain management for patients without resorting to opioids when a non-opioid alternative would suffice. It provides pertinent clinical information to the dentist, including point-of-care access to the Prescription Drug Monitoring Program.
  Interventions: Other: Clinical Decision Support
- Clinical Decision Support + Education (Experimental): Patient education regarding pain management before and after dental extraction, including information about the risks and benefits of various strategies.
  Interventions: Other: Clinical Decision Support; Other: Patient education

INTERVENTIONS:
Other: Clinical Decision Support — A clinical decision support system designed to assist dentists in providing optimal pain management for patients without resorting to opioids when a non-opioid alternative would suffice. It provides pertinent clinical information to the dentist, including point-of-care access to the Prescription Drug Monitoring Program.
  Arms: Clinical Decision Support; Clinical Decision Support + Education
Other: Patient education — Patient education regarding pain management before and after dental extraction, including information about the risks and benefits of various strategies.
  Arms: Clinical Decision Support + Education

SUMMARY:
The overarching goal of this project is to de-implement the reliance on opioid analgesics and to implement reliance on non-opioid analgesics to manage postoperative pain following dental extractions. Using a prospective, provider-level, 3-arm cluster randomized trial design, the investigators will compare different strategies to reduce the reliance on opioids and increase the use of alternative pain management approaches utilizing information support tools aimed at both providers and their patients.

DETAILED DESCRIPTION:
The primary objective of this project is to de-implement the use of opioid analgesics for the management of postoperative pain following dental extractions and to implement effective alternative pain management. The investigators propose a cluster-randomized trial design in which dental practitioners will be randomly assigned to 1 of 3 conditions involving different implementation strategies. The first condition, Standard Practice, will serve as a control condition. The second condition will implement a clinical decision support (CDS) tool that will extract patient history and interface with the state prescription drug monitoring program to provide personalized recommendations for analgesic prescribing and offer language for discussing optimal, evidence-based non-opioid pain management with dental extraction patients. The third condition will involve an enhanced version of the CDS (CDS-E) that will also include information regarding optimal, evidence-based, non-opioid pain management delivered directly to the patient both before and following the dental extraction visit. The investigators will examine opioid and non-opioid prescribing data from the electronic health record across study arms as well as other provider- and patient-focused outcomes using mixed methods.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Have a dental extraction of a permanent teeth performed by an eligible HealthPartners provider during the intervention period

Exclusion Criteria:

* Patients who have opted out of research at HealthPartners
* Meet above age criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5722 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Brad Rindal, DDS, Principal Investigator — HealthPartners Institute; Shannon G. Mitchell, PhD, Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- HealthPartners Dental Group, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data outputs: patient survey data, Electronic Health Record (EHR) study data
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Release of de-identified datasets and accompanying technical resources used for specific publications will occur within 6 months of the online publication date.
Access Criteria: Data will be stored at HealthPartners Institute by the project co-principal investigator/site lead and statistician. Study publications will note the method for requesting the study data and technical materials. The study statistician will provide data and accompanying files in an archived zip format to requesters via email. Data will not be stored in a public repository.

REFERENCES:
- [Background] Rindal DB, Asche SE, Gryczynski J, Kane SM, Truitt AR, Shea TL, Ziegenfuss JY, Schwartz RP, Worley DC, Mitchell SG. De-Implementing Opioid Use and Implementing Optimal Pain Management Following Dental Extractions (DIODE): Protocol for a Cluster Randomized Trial. JMIR Res Protoc. 2021 Apr 12;10(4):e24342. doi: 10.2196/24342. PMID 33843594
- [Background] Mitchell SG, Truitt AR, Davin LM, Rindal DB. Pain management after third molar extractions in adolescents: a qualitative study. BMC Pediatr. 2022 Apr 7;22(1):184. doi: 10.1186/s12887-022-03261-x. PMID 35392856
- [Background] Rindal DB, Asche SE, Kane S, Truitt AR, Worley DC, Davin LM, Gryczynski J, Mitchell SG. Patient, Provider Type, and Procedure Type Factors Associated with Opioid Prescribing by Dentists in a Health Care System. J Pain Res. 2021 Oct 20;14:3309-3319. doi: 10.2147/JPR.S330598. eCollection 2021. PMID 34707399
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Derived] Mitchell SG, Gryczynski J, Worley DC, Asche SE, Truitt AR, Rindal DB. Barriers to dental providers' use of a clinical decision support tool for pain management following tooth extractions. Implement Res Pract. 2025 Feb 9;6:26334895251319810. doi: 10.1177/26334895251319810. eCollection 2025 Jan-Dec. PMID 39931509
- [Derived] Rindal DB, Pasumarthi DP, Thirumalai V, Truitt AR, Asche SE, Worley DC, Kane SM, Gryczynski J, Mitchell SG. Clinical Decision Support to Reduce Opioid Prescriptions for Dental Extractions using SMART on FHIR: Implementation Report. JMIR Med Inform. 2023 Nov 7;11:e45636. doi: 10.2196/45636. PMID 37934572
- [Derived] Gryczynski J, Mitchell SG, Asche SE, Truitt AR, Worley DC, Rindal DB. De-Implementing Opioids for Dental Extractions (DIODE): a multi-clinic, cluster-randomized trial of clinical decision support strategies in dentistry. Implement Sci. 2023 Feb 10;18(1):5. doi: 10.1186/s13012-023-01262-7. PMID 36765414
- [Derived] Rindal DB, Gryczynski J, Asche SE, Truitt AR, Kane SM, Worley DC, Mitchell SG. De-implementing opioid prescribing in a dental group practice: Lessons learned. Community Dent Oral Epidemiol. 2023 Feb;51(1):139-142. doi: 10.1111/cdoe.12820. Epub 2023 Feb 8. PMID 36753410
- Available data/document: Study Protocol — https://www.researchprotocols.org/2021/4/e24342

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Dentists
Groups:
- Standard Practice: Standard Practice: The patients in this arm were part of usual care with their dental provider.
Period: Overall Study
Arm/Group | Standard Practice | Clinical Decision Support | Clinical Decision Support + Education
Started | 1739; 17 Dentists | 2297; 16 Dentists | 1686; 17 Dentists
Completed | 1720; 16 Dentists | 2269; 14 Dentists | 1660; 13 Dentists
Not Completed | 19; 1 Dentists | 28; 2 Dentists | 26; 4 Dentists
Not completed — refused EHR permission | 19 | 28 | 23
Not completed — patients tied to a provider who retired | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: 73 participants declined use of their EHR data
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Practice | Clinical Decision Support | Clinical Decision Support + Education | Total
Number analyzed (Participants) | 1720 | 2269 | 1660 | 5649
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 115 | 151 | 89 | 355
  Between 18 and 65 years | 1290 | 1598 | 1136 | 4024
  >=65 years | 315 | 520 | 435 | 1270
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (19.4) | 46.6 (20.6) | 49.7 (20.0) | 47.2 (20.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1019 | 1284 | 937 | 3240
  Male | 701 | 985 | 723 | 2409
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 113 | 71 | 275
  Not Hispanic or Latino | 1274 | 1479 | 1073 | 3826
  Unknown or Not Reported | 355 | 677 | 516 | 1548
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13 | 17 | 11 | 41
  Asian | 142 | 183 | 132 | 457
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 3 | 7
  Black or African American | 324 | 421 | 284 | 1029
  White | 953 | 1217 | 950 | 3120
  More than one race | 14 | 29 | 10 | 53
  Unknown or Not Reported | 272 | 400 | 270 | 942

OUTCOME MEASURES:

1. Primary Outcome: Opioid Prescribing at the Extraction Encounter
Description: Number of participants prescribed an opioid.
Time Frame: At the extraction encounter
Population: 73 participants declined use of their EHR data
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Practice | Clinical Decision Support | Clinical Decision Support + Education
Number analyzed (Participants) | 1720 | 2269 | 1660
Participants | 443 | 643 | 418
Statistical Analysis 1: Comparison: Standard Practice vs Clinical Decision Support; Test type: Superiority; p = .08, Mixed Models Analysis; Odds Ratio (OR) = 1.29, 97.5% CI 2-sided [.93 to 1.80]
Statistical Analysis 2: Comparison: Standard Practice vs Clinical Decision Support + Education; Test type: Superiority; p = .18, Mixed Models Analysis; Odds Ratio (OR) = 1.24, 97.5% CI 2-sided [.86 to 1.79]

2. Secondary Outcome: Exclusive Non-opioid Prescribing or Recommendations at the Extraction Encounter
Description: Number of participants prescribed or recommended non-opioid analgesics (ibuprofen, naproxen, aspirin, or acetaminophen) and did not prescribe opioids (at the time of the extraction encounter).
Time Frame: At the extraction encounter
Population: 73 participants declined use of their EHR data
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Practice | Clinical Decision Support | Clinical Decision Support + Education
Number analyzed (Participants) | 1720 | 2269 | 1660
Participants | 714 | 888 | 566
Statistical Analysis 1: Comparison: Standard Practice vs Clinical Decision Support; Test type: Superiority; p = .71, Mixed Models Analysis; Odds Ratio (OR) = 1.37, 97.5% CI 2-sided [.20 to 9.44]
Statistical Analysis 2: Comparison: Standard Practice vs Clinical Decision Support + Education; Test type: Superiority; p = .62, Mixed Models Analysis; Odds Ratio (OR) = 1.53, 97.5% CI 2-sided [.21 to 11.00]

3. Secondary Outcome: Compare the Study Arm Differences in Shared Decision-making
Description: The CollaboRATE scale measures shared decision making and consists of the mean of three items, each rated on a 0 ("no effort was made") to 4 ("every effort was made") scale. The possible range for the composite score is 0-4, with a higher score on the scale indicating that more shared decision-making occurred.
Time Frame: 3-6 days after the extraction encounter
Population: The information for this endpoint is based on a survey of patients and was offered to a sample of patients among the 5722 in the larger study.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard Practice | Clinical Decision Support | Clinical Decision Support + Education
Number analyzed (Participants) | 157 | 199 | 136
score on a scale | 3.3 [3.2 to 3.5] | 3.3 [3.2 to 3.4] | 3.3 [3.2 to 3.4]
Statistical Analysis 1: Comparison: Standard Practice vs Clinical Decision Support; Test type: Superiority; p = .38, Mixed Models Analysis; Median Difference (Net) = -0.07, 95% CI 2-sided [-0.26 to .12]
Statistical Analysis 2: Comparison: Standard Practice vs Clinical Decision Support + Education; Test type: Superiority; p = .70, Mixed Models Analysis; Median Difference (Net) = -0.03, 95% CI 2-sided [-0.24 to .17]

4. Secondary Outcome: Compare the Study Arm Differences in Patient Experiences of Post-extraction Pain
Description: Study arm comparison of the average patient-reported pain 3 days following the extraction encounter. (Numeric Rating Scale, 0 'no pain at all' - 10 'worst pain imaginable')
Time Frame: 3-6 days after the extraction encounter
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Standard Practice | Clinical Decision Support | Clinical Decision Support + Education
Number analyzed (Participants) | 157 | 199 | 136
score on a scale | 3.8 [3.3 to 4.3] | 3.7 [3.2 to 4.1] | 3.5 [3.0 to 4.0]
Statistical Analysis 1: Comparison: Standard Practice vs Clinical Decision Support; Test type: Superiority; p = .65, Mixed Models Analysis; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.79 to .50]
Statistical Analysis 2: Comparison: Standard Practice vs Clinical Decision Support + Education; Test type: Superiority; p = .41, Mixed Models Analysis; Mean Difference (Net) = -0.29, 95% CI 2-sided [-0.99 to .41]

ADVERSE EVENTS:
Time Frame: Through 7 days following the extraction encounter.
Description: We are following the standard definition. In addition, potential Adverse Events included subsequent opioid prescribing assessed through Electronic Health Record (EHR) data.
Arm/Group | Standard Practice | Clinical Decision Support | Clinical Decision Support + Education
All-Cause Mortality (participants affected / at risk) | 0/1720 | 0/2269 | 0/1660
Serious Adverse Events (participants affected / at risk) | 0/1720 | 0/2269 | 0/1660
Other Adverse Events (participants affected / at risk) | 0/1720 | 1/2269 | 0/1660
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Practice (N=1720) | Clinical Decision Support (N=2269) | Clinical Decision Support + Education (N=1660)
Pain at site (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — No opioid prescribed at extraction visit, same day call to care line resulted in prescription.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03584789/Prot_SAP_000.pdf